CLINICAL TRIAL: NCT03724461
Title: Effects of Resistance Training With High vs. Light-moderate Loads on Muscle-tendon Function in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); Biomedical Research Networking Center on Frailty and Healthy Aging (CIBERFES) (Unknown)
Responsible Party: Principal Investigator, Luis M. Alegre, Associate Professor, University of Castilla-La Mancha
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: DEP2015-69386-R
Record Dates: First submitted 2018-09-18; First posted 2018-10-30 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Aging; Sarcopenia; Frail Elderly Syndrome
Keywords: resistance training; sarcopenia; hypertrophy; tendon; frailty; ageing
MeSH Terms: conditions — Sarcopenia; Hypertrophy; Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- High intensity vs Control (12 weeks) (Active Comparator): 8 weeks of baseline period plus an exercise program where one leg undergoes High Intensity resistance training (12 weeks) and the other leg is established as control.
  Interventions: Behavioral: High Intensity resistance training (12 weeks); Behavioral: Control (12 weeks)
- Light intensity vs Control (12 weeks) (Active Comparator): 8 weeks of baseline period plus an exercise program where one leg undergoes light-moderate intensity resistance training (12 weeks) and the other leg is established as control.
  Interventions: Behavioral: Light-moderate intensity resistance training (12 weeks); Behavioral: Control (12 weeks)
- High vs Light intensity (12 weeks) (Experimental): 8 weeks of baseline period plus an exercise program where one leg undergoes High Intensity resistance training (12 weeks) and the other leg undergoes light-moderate intensity resistance training.
  Interventions: Behavioral: High Intensity resistance training (12 weeks); Behavioral: Light-moderate intensity resistance training (12 weeks)
- High intensity (Acute) (Experimental): Analysis of the effects of one High Intensity resistance training session, with a crossover design.
  Interventions: Behavioral: One High Intensity resistance training session
- Light intensity (Acute) (Experimental): Analysis of the effects of one Light-moderate Intensity resistance training session, with a crossover design.
  Interventions: Behavioral: One Light-moderate intensity resistance training session

INTERVENTIONS:
Behavioral: High Intensity resistance training (12 weeks) — High intensity resistance training (80% of 1 repetition maximum), 2 d/wk (Longitudinal)
  Other Names: HIT
  Arms: High intensity vs Control (12 weeks); High vs Light intensity (12 weeks)
Behavioral: Light-moderate intensity resistance training (12 weeks) — Light-moderate intensity resistance training (40% of 1 repetition maximum), 2 d/wk (Longitudinal)
  Other Names: LIT
  Arms: High vs Light intensity (12 weeks); Light intensity vs Control (12 weeks)
Behavioral: Control (12 weeks) — No resistance training during the intervention period.
  Other Names: CON
  Arms: High intensity vs Control (12 weeks); Light intensity vs Control (12 weeks)
Behavioral: One High Intensity resistance training session — High intensity resistance training, 1 training session
  Other Names: HIT (Acute)
  Arms: High intensity (Acute)
Behavioral: One Light-moderate intensity resistance training session — Light-moderate intensity resistance training, 1 training session
  Other Names: LIT (Acute)
  Arms: Light intensity (Acute)

SUMMARY:
There are no unbiased studies that have analyzed the effects of resistance training with traditional, heavy versus light-moderate loads on muscle, tendon and bone in elderly people.

The purpose of the present study is to assess the effects on muscle mass and function, tendon and bone of two different training intensities, light-moderate vs. heavy load, in people older than 65 years old.

The study will be carried out with a randomized controlled design. Participants will perform single training sessions and a 12-wk dynamic resistance training program on the knee extensors with different training intensities on each leg. One leg will train with heavy loads and the other one will train with light-moderate loads, but matching the load x repetitions performed by the contralateral side.

DETAILED DESCRIPTION:
The decline in muscle function provoked by the aging process and frailty are directly related to decreases in mobility and the ability to perform the so called "daily life activities". Resistance training is especially useful at this stage, given that it is an effective and widely applicable intervention to control and revert sarcopenia, and the deterioration of tendon and bone function. Despite of the effectiveness of heavy load resistance training, a controversy has arisen in the last years about the effects of lower load resistance training programs to achieve similar adaptations. This is because most of the studies that have compared light-moderate versus heavy load programs did not control the differences in total training load, measured as the overall mechanical work performed during the training program. Therefore, there are no unbiased studies that have analyzed the effects of resistance training with traditional, heavy versus light-moderate loads on muscle, tendon and bone in elderly people.

The purpose of the present study is to assess the effects on muscle mass and function, tendon and bone of two different training intensities, light-moderate vs. heavy load, in people older than 65 years old.

The studies will be carried out with a crossover (acute training sessions) and randomized controlled design (longitudinal training intervention). Participants will perform single training sessions with each resistance training intensity and a 12-wk dynamic resistance training program on the knee extensors with different training intensities on each leg. One leg will train with heavy loads and the other one will train with light-moderate loads, but matching the load x repetitions performed by the contralateral side. Muscle adaptations (EMG, muscle size and architecture), tendon mechanical properties, bone mineral density, blood parameters and life quality will be analyzed before and after the cessation of the training program.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older,
* non-institutionalized
* passed physical examination including physical function assessment (no frailty status; SPPB >7 points)

Exclusion Criteria:

* Neurological, musculoskeletal, or other disorder that would preclude completing resistance training and all performance tests
* Uncontrolled hypertension, unstable or exercise-induced angina pectoris or myocardial ischemia or any other medical condition that would interfere with testing or increase one's risk of complications during exercise.
* History of regular resistance exercise during the previous 3 years
* Knee prosthesis

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Acute change in muscle size (cross sectional area, cm2) | Change from baseline at 5 minutes after a training session
  Ultrasound-based determination quadriceps muscle size and architecture.
Change in muscle size (cross sectional area, cm2) | Change from baseline to week 12
  Ultrasound-based determination quadriceps muscle size and architecture.
Acute change in muscle function (N) | Change from baseline at 5 minutes after a training session
  Force-velocity profile of the single-leg press exercise
Change in muscle function (N) | Change from baseline to week 12
  Force-velocity profile of the single-leg press exercise

SECONDARY OUTCOMES:
Change in patellar tendon stiffness (N/mm) | Change from baseline to week 12
  Ultrasound and force-based measures of tendon mechanical properties.
Acute change in patellar tendon stiffness (N/mm) | Change from baseline at 5 minutes after a training session
  Ultrasound and force-based measures of tendon mechanical properties.
Change in muscle mass (kg) | Change from baseline to week 12
  Lean mass determined by Dual energy X-ray absorptiometry
Change in bone mass (g) | Change from baseline to week 12
  Bone mineral content determined by Dual energy X-ray absorptiometry
Acute change in muscle excitation (mV) | Change from baseline at 5 minutes after a training session
  Electromyographic activity of the knee extensor and flexor muscles during strength assessment and training
Change in muscle excitation (mV) | Change from baseline to week 12
  Electromyographic activity of the knee extensor and flexor muscles during strength assessment and training
Change in physical function | Change from baseline to week 12
  Short Physical Performance Battery
Blood analysis: Acute change in oxidative stress | Change from baseline at 5 minutes after a training session
  Carbonyl proteins (plasma concentration)
Blood analysis: Change in oxidative stress | Change from baseline to week 12
  Carbonyl proteins (plasma concentration)
Blood analysis: Acute change in Inflammation | Change from baseline at 5 minutes after a training session (Acute)
  Interleukin 6, Tumoral necrosis factor Alpha, C reactive protein (plasma concentration)
Blood analysis: Change in inflammation | Change from baseline to week 12
  Interleukin 6, Tumoral necrosis factor Alpha, C reactive protein (plasma concentration)
Blood analysis: Acute change in anabolic processes | Change from baseline at 5 minutes after a training session
  Testosterone, growth hormone, Insulin growth factor-1 (plasma concentration)
Blood analysis: Change in anabolic processes | Change from baseline to week 12
  Testosterone, growth hormone, Insulin growth factor-1 (plasma concentration)
Blood analysis: Acute change in catabolic processes | Change from baseline at 5 minutes after a training session
  Cortisol, Creatin kinase (plasma concentration)
Blood analysis: Change in catabolic processes | Change from baseline to week 12
  Cortisol, Creatin kinase (plasma concentration)

CONTACTS AND LOCATIONS:
Overall Officials: Luis M. Alegre, PhD, Principal Investigator — Associate Professor
Locations (1):
- Universidad de Castilla-La Mancha, Laboratorio de Actividad Física y Función Muscular. Campus de la Fábrica de Armas. Avda. Carlos III s/n, Toledo, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rodriguez-Lopez C, Alcazar J, Sanchez-Martin C, Baltasar-Fernandez I, Ara I, Csapo R, Alegre LM. Contralateral Adaptations After Unilateral Power Training in Older Adults: The Effect of Intensity of Load. Scand J Med Sci Sports. 2025 Nov;35(11):e70165. doi: 10.1111/sms.70165. PMID 41222282
- [Derived] Rodriguez-Lopez C, Alcazar J, Losa-Reyna J, Martin-Espinosa NM, Baltasar-Fernandez I, Ara I, Csapo R, Alegre LM. Effects of Power-Oriented Resistance Training With Heavy vs. Light Loads on Muscle-Tendon Function in Older Adults: A Study Protocol for a Randomized Controlled Trial. Front Physiol. 2021 Feb 18;12:635094. doi: 10.3389/fphys.2021.635094. eCollection 2021. PMID 33679447
- [Derived] Rodriguez-Lopez C, Alcazar J, Sanchez-Martin C, Ara I, Csapo R, Alegre LM. Mechanical Characteristics of Heavy vs. Light Load Ballistic Resistance Training in Older Adults. J Strength Cond Res. 2022 Aug 1;36(8):2094-2101. doi: 10.1519/JSC.0000000000003826. Epub 2020 Sep 16. PMID 32947572